CLINICAL TRIAL: NCT06127082
Title: Left Cardiac Chambers Size in Obese Individuals and Its Relation to BMI and Waist
Brief Title: Left Cardiac Chambers Size in Obese Individuals and Its Relation to BMI and Waist Circumference
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Baha Elia, Resident doctor at internal medicine department, Assiut University
Other Study IDs: The effect of obesity on heart
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echocardiography — Do echocardiography to obese patient

SUMMARY:
Aim of study:

To determine if there is relation between left cardiac chambers size ,BMI and waist circumference in obese individuals.

1. Primary outcomes:

   -To determine if there is relation between left cardiac chambers size ,BMI and waist circumference in obese individuals.
2. Secondary outcomes:

   * To determine the effect of obesity on heart health in obese individuals.

DETAILED DESCRIPTION:
Body mass index and waist circumference are important measurements of our bodies as they can affect our health.The person is obese if he has BMI equal 30 or higher.Increased risk of obesity related disease occurs in men with waist circumference equal 102 cm or more and woman with waist circumference equals 88 cm or more. increasing BMI and waist circumference can increase risk of type 2 diabetes mellitus ,hypertension ,cardiovascular disease and cerebrovascular accidents.There are many diseases that can affect left cardiac chambers size like aortic, mitral valvediseases,hypertension and atherosclerosis.Screening of patients heart by echocardiography allow us to detect changes in the muscle of heart and this allow doctors to put treatment plan to patient to prevent heart health from deterioration. In this study the investigators want to know if there an association between left cardiac chambers size ,BMI and waist circumference in obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* 1-Patient age 18 years old or above. 2-Patient BMI 30kg/m2 or higher . 3-Patient waist circumference in men 102cm or more and in women 88cm or more. 4-Obese patient with comorbidities (e.g DM,HTN).

Exclusion Criteria:

* 1-Patient age 18 years old. 2-Patient BMI less than 30 kg/m2. 3-Patient waist circumference in men less than 102cm and in women less than 88cm.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - 1-Patient age 18 years old or above. 2-Patient BMI 30kg/m2 or higher . 3-Patient waist circumference in men 102cm or more and in women 88cm or more. 4-Obese patient with comorbidities (e.g DM,HTN).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
To determine if there is correlation between left cardiac chambers size in mm ,BMI in kg/m^2 and waist circumference in cm in obese individuals | Baseline
  effect of obesity on left cardiac chambers size

SECONDARY OUTCOMES:
To determine the effect of obesity on heart health in obese individuals. | Baseline
  effect of obesity on left cardiac chambers size

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Anwar, professor, Study Director — Assiut University

REFERENCES:
- [Background] Moukarzel J, Guevara E, Casciaro ME, Guilenea FN, Pascaner AF, Craiem D. Echocardiographic Measurements of Left Heart Chamber Size in a Large Cohort of Subjects: Comparison of Body Surface Area and Height Indexing to Account for Effects of Obesity. J Am Soc Echocardiogr. 2022 Nov;35(11):1159-1167.e2. doi: 10.1016/j.echo.2022.08.001. Epub 2022 Aug 8. PMID 35953008